CLINICAL TRIAL: NCT05503433
Title: Effect of Maternal Cortisol Levels on Fetal Heart Rate Patterns
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Other Study IDs: FKH Parameters
Record Dates: First submitted 2022-08-08; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Stress; Cortisol; Hypersecretion; Fetal Heart Rate Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: This study was designed to determine whether maternal cortisol levels affect fetal heart rate (FHR) patterns at third trimester.

Design: Cross-sectional descriptive study. Setting: Prenatal wards of 1 public maternity services in Istanbul, Turkey. Participants: This study included 400 nulliparous pregnant women with uncomplicated pregnancies with a single fetus, between October 2022 and December 2022.

Measurements and Findings:

The minimum sample size required in the study was decided by power analysis. Effect size in the calculation: 0.35, type 1 error rate (α)=0.05, power of the study (1- β) 0.95 (Type II error=0.05) taken as. Accordingly, the minimum number of samples to be reached was calculated as 356 in total, and it was aimed to reach 392 samples, taking into account the 10% risk of loss.

Research data will collect with the Data Collection Form. Noise level will measure with the Personal Noise Dosimeter. The FHR data will collect using a cardiotocograph. Saliva cortisol will measure by a microplate reader with commercially available kit based on ELISA.

DETAILED DESCRIPTION:
Pregnancy is associated with psychological stress for many reasons such as physiological, social and emotional changes. In the literature, it is thought that the stress experienced in the prenatal period may affect maternal and fetal health primarily and secondarily. Primary factors; It is the direct effect of increasing stress during pregnancy on biological systems (increasing stress hormones on the body). Secondary factors are; It is an indirect effect on maternal and fetal health as a result of unhealthy behaviors such as substance use and not going to prenatal check-ups in pregnant women who experience stress symptoms. In both ways, stress is associated with adverse maternal, fetal, neonatal and long-term outcomes. Prenatal stress; It is reported to increase the risk of hypertensive diseases, placental abnormalities, increased uterine, arterial resistance, spontaneous abortion, antenatal bleeding, preterm labor, difficult labor, operative deliveries, postpartum depression, intrauterine growth retardation, low APGAR Score, low birth weight and fetal death. Along with these, maternal anxiety seemed to affect the duration and variability of the FHR, with prolonged accelerations often fused into sustained tachycardia. A further paper reported that the children of women who were highly anxious during pregnancy were more likely to be hyperactive, more likely to show attention deficit, and more likely to exhibit difficult behavior and aggression compared with children from low anxiety mothers.

Fetal heart rate (FHR) monitoring is the primary clinical technique for assessing fetal well-being and is one of the most useful techniques for investigating fetal neurodevelopment. In addition, FHR acceleration (defined as > 15 beats/min from baseline) is associated with fetal movement (fetal reactivity) and has been found to have a high association with fetal well-being.

Before 24 weeks gestation, fetal reactivity is rare, and it would seem that the appearance of FHR reactivity is related to maturation of the central nervous system (CNS), which occurs at the beginning of the third trimester. In research which conducted in 2010, found that fetuses of women who had a cortisol increase following an arithmetic task versus those who did not, had higher resting (HR) and less short-term HR variability (HRV) 20 min after the stressor task ended. There was a trend finding for participants who had a cortisol increase to report higher levels of life stress. In other research, higher resting maternal cortisol during the 3rd trimester was associated with greater amplitude and amount (time spent) of fetal movement during a 50-min observation period. The aim of the present study was to determine determine whether maternal cortisol levels affect fetal heart rate (FHR) patterns.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research,
* Over 18 years old,
* Literate,
* Speaks Turkish,
* In the third trimester of pregnancy,
* Having a healthy pregnancy,
* No adrenal insufficiency,
* No problems with hearing,
* No psychiatric diagnosis during or before pregnancy,
* No history of infertility,
* Coming to routine pregnancy and NST control,
* Have not had any food or drink for at least two hours before the procedure,
* Nulliparous pregnant women without contractions were included.

Exclusion Criteria:

* Pregnant women whose contractions are detected while the NST procedure is in progress,
* Pregnant women with deceleration detected in the NST procedure were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nulliparous pregnant women
Study Population: In all patients, well-being and growth of the fetus should be normal and amniotic fluids were also normal.
Sampling Method: Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Maternal cortisol level of the pregnant women | 01.02.2021-01.10.2021
  About 5 ml of maternal saliva for cortisol measurements will collect at 08:00 -10:00 h and store at -80 °C until analysis. Saliva cortisol will measure by a microplate reader (Thermo Scientific Multiskan FC, 2011-06, USA) with commercially available kit based on ELISA (Human Salivary Cortisol ELISA kit-DRG international, Inc., USA, Cat Num:slv-2930).

SECONDARY OUTCOMES:
Fetal heart rate measurement | 01.02.2021-01.10.2021
  The Fetal Heart Rate data will collect using a cardiotocograph (Philips Avalon FM20).

REFERENCES:
- [Derived] Turan A, Kaya C. Effect of maternal cortisol levels on fetal heart rate patterns in primiparous pregnant women in the third trimester. Rev Assoc Med Bras (1992). 2023 May 19;69(5):e20221610. doi: 10.1590/1806-9282.20221610. eCollection 2023. PMID 37222328